CLINICAL TRIAL: NCT02331056
Title: Could the Stroke Volume Variation Predict a Fluid Responsiveness in Thoracotomy?
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Associate professor, Samsung Medical Center
Other Study IDs: 2014-06-053-002
Record Dates: First submitted 2014-12-15; First posted 2015-01-05 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Neoplasm; Pulmonary Tuberculosis
Keywords: Stroke volume variation; fluid responsiveness; One-lung ventilation; thoracotomy
MeSH Terms: conditions — Lung Neoplasms; Tuberculosis, Pulmonary | interventions — Thoracotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- thoracoscopic pulmonary lobectomy: to observe a fluid responsiveness in patients who receives scheduled thoracoscopic pulmonary lobectomy
  Interventions: Other: fluid loading; Procedure: thoracoscopic pulmonary lobectomy
- open pulmonary lobectomy(thoracotomy): to observe a fluid responsiveness in patients who receives scheduled open pulmonary lobectomy(thoracotomy)
  Interventions: Other: fluid loading; Procedure: thoracotomy

INTERVENTIONS:
Other: fluid loading — Fluid loading at defined period
  * 500ml colloid solution infusion at 20min after thorax open for 30min. 500ml colloid administration is a kind of routine procedure during pulmonary lobectomy in our hospital. We just control the fluid loading timing for hemodynamic parameter records.
Procedure: thoracoscopic pulmonary lobectomy — the patient group for scheduled thoracoscopic pulmonary lobectomy
  Groups: thoracoscopic pulmonary lobectomy
Procedure: thoracotomy — the patient group for scheduled open pulmonary lobectomy
  Groups: open pulmonary lobectomy(thoracotomy)

SUMMARY:
There are some risks of pulmonary edema in patients undergoing pulmonary lobectomy with one lung ventilation. The overloading of fluid administration could be related to the development of pulmonary edema in patents after thoracic surgery. But fluid restriction may cause major organ hypoperfusion during the surgery. The purpose of this study is to evaluate the ability of stroke volume variation as an indicator for a fluid responsiveness in patient who receives pulmonary lobectomy via thoracotomy.

DETAILED DESCRIPTION:
Perioperative fluid management during thoracic surgery is a significantly important, because it is quite difficult to prevent pulmonary edema due to the fluid overload and compromise perfusion of vital organ. So, it is essential to maintain optimal organ perfusion by appropriate fluid management during thoracic surgery. Stroke volume variation (SVV) is derived from pulse contour analysis and it is known that SVV ≥12~15% correlate with fluid responsiveness, defined as a significant increase in cardiac output with fluid loading, dung two-lung ventilation. It is a parameter derived from changes in stroke volume (SV) that is according to the heart-lung interaction during mechanical ventilation. positive pressure ventilation induces cyclic changes in left ventricular SV that are related mainly to the expiratory decrease in right ventricular filling and ejection. This is a reflected by variations in the SV. However both ventilator issues, such as tidal volume, PEEP, chest and lung condition, and the cardiovascular condition, such as heart rate, rhythm, ventricular function, cardiac afterload, arterial compliance may affect SVV. Recently some studies reported that SVV could predict fluid responsiveness in mechanically ventilated patients under various conditions. But it is still unclear whether SVV could predict fluid responsiveness during one lung ventilation with the chest open via a thoracotomy. During one-lung ventilation, the shunted blood flow through the non-ventilated-lung dose not contribute to the generation of SVV. And with the chest opening by thoracotomy, the pressure generated by ventilator would not be transmitted to the pulmonary vessels but rather to the atmosphere. So, the purpose of this study is to evaluate the ability of SVV as an indicator a fluid responsiveness particularly in patients undergoing one-lung ventilation with thoracotomy and to found the optimal threshold value of SVV for fluid management during thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients scheduled for pulmonary lobectomy with one lung ventilation by lung cancer, nodule, or pulmonary tuberculosis under thoracoscopy or thoracotomy in our hospital

Exclusion Criteria:

* The patients with known cardiac disease include arrythmia
* American society of anesthesia physical status III, IV, V

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients scheduled for pulmonary lobectomy with one lung ventilation by lung cancer, nodule, or pulmonary tuberculosis under thoracoscopy or thoracotomy in our hospital were included.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in SVV, SVI after fluid loading | 20min after thorax open and immediate after fluid loading for 30min
  we are going to measure the SVV, SVI before and after fluid loading. Fluid responders were defined as patients demonstrating an increase in SVI ≥ 10% and non-responders as patients whose SVI changed < 10%. Receiver operating characteristic (ROC) curves were generated for SVV of each group (responders and non responders). Threshold value of SVV was determined by considering values that yielded the greatest sensitivity and specificity from ROC curve

OTHER OUTCOMES:
Number of Participants with Adverse Events (pulmonary complication) | participants will be followed for the duration of hospital stay, an expected average of 1 week
  after surgery check chest x-ray It's the routine follow up after lobectomy.
Number of Participants with Adverse Events (compromise perfusion of vital organ ) | participants will be followed for the duration of hospital stay, an expected average of 1 week
  check perioperative urine output, and check post op serum creatine

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

REFERENCES:
- [Derived] Jeong DM, Ahn HJ, Park HW, Yang M, Kim JA, Park J. Stroke Volume Variation and Pulse Pressure Variation Are Not Useful for Predicting Fluid Responsiveness in Thoracic Surgery. Anesth Analg. 2017 Oct;125(4):1158-1165. doi: 10.1213/ANE.0000000000002056. PMID 28504996